CLINICAL TRIAL: NCT05712317
Title: Evaluation of the Effectiveness of Regular Training in the ExerCube - A Randomized Controlled Trial
Brief Title: The Effectiveness of an Exergame-based Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-03-00006
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Blood Pressure; Physical Inactivity
Keywords: Exergaming; Blood pressure; Endurance performance; Pulse wave analysis; Exercise
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame Intervention (Experimental): 8-week exergame-based intervention consisting of 3 sessions per week lasting between 20-40 Minutes. The intervention will consist of playing the game Sphery racer in the exergame called ExerCube.
  Interventions: Behavioral: Exergame Intervention
- Moderate-intensity endurance exercise (Active Comparator): 8-week moderate-intensity endurance exercise consisting of 3 sessions per week lasting between 20-40 minutes. The intervention will consist of a running exercise on a treadmill or riding on a bicycle ergometer.
  Interventions: Behavioral: Moderate-intensity endurance exercise

INTERVENTIONS:
Behavioral: Exergame Intervention — 8-week exergame-based intervention 3x per week
  Arms: Exergame Intervention
Behavioral: Moderate-intensity endurance exercise — 8-week moderate-intensity endurance exercise 3x per week
  Arms: Moderate-intensity endurance exercise

SUMMARY:
This randomized control trial aims to compare the effects of a regular exergame-based intervention and a regular moderate-intensity endurance exercise in healthy individuals. The main questions it aims to answer are:

• Is regular exergame-based training an effective intervention to improve different health and performance parameters in healthy adults? Can the exergaming intervention improve health and performance parameters similar to a moderate-intensity endurance exercise intervention? Throughout the intervention period (8 weeks), participants will participate in regular training sessions (3x/week) in an exergame called the ExerCube.

Researchers will compare the effects to a control group who participates in regular (3x/week) moderate-intensity endurance exercise to see if the exergaming intervention induces similar effects on health and performance parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male adults
* Aged 18-60 years
* Free from acute and chronic diseases
* Free from movement restrictions or injuries to the musculoskeletal system
* Provided written informed consent

Exclusion Criteria:

* Underlying health condition that could compromise the safety of the physical exercise
* Were taking cardiovascular medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in maximum oxygen consumption at week 8 | Baseline and week 8
  Maximum oxygen consumption will be obtained during a cardiopulmonary exercise test on a bicycle ergometer using a validated metabolic cart.

SECONDARY OUTCOMES:
Changes from baseline in pulse wave velocity at week 8 | Baseline and week 8
  Pulse wave velocity will be obtained non-invasively using a clinically validated device for hemodynamic measurements. After a 10 min supine rest, a minimum of two readings will be performed on the right upper arm using customized arm cuffs.
Changes from baseline in systolic blood pressure at week 8 | Baseline and week 8
  Systolic blood pressure will be obtained non-invasively using a clinically validated device for hemodynamic measurements. After a 10 min supine rest, a minimum of two readings will be performed on the right upper arm using customized arm cuffs.
Changes from baseline in diastolic blood pressure at week 8 | Baseline and week 8
  Diastolic blood pressure will be obtained non-invasively using a clinically validated device for hemodynamic measurements. After a 10 min supine rest, a minimum of two readings will be performed on the right upper arm using customized arm cuffs.

OTHER OUTCOMES:
Changes from baseline in body mass index at week 8 | Baseline and week 8
  Height will be measured barefoot with a stadiometer to the nearest 0.5 cm. Body mass will be measured using a scale. Body mass index will be calculated as a function of weight in kilogram and height in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Ketelhut, Dr., Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available upon reasonable request from the principal investigator.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the intervention is over and all data is obtained.
Access Criteria: Reasonable request .